CLINICAL TRIAL: NCT06340087
Title: Einfluss Des Süßmodulierenden Polyphenols Hesperetin in Kombination Mit Saccharose Auf Die Blutglukose-Regulierung Und Energieaufnahme in Abhängigkeit Der Süßwahrnehmung Teil 2
Brief Title: Impact Hesperetin in Combination with Sucrose on Blood Glucose Regulation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Barbara Lieder, Professor and Vice Chair Department of Physiological Chemistry, University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 706014-3
Record Dates: First submitted 2024-03-24; First posted 2024-04-01 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Blood Glucose Fluctuations; Hunger
MeSH Terms: interventions — Sucrose; Dietary Sucrose

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 10% Sucrose (Experimental): 10% (w/v) sucrose in water
  Interventions: Other: 10% Sucrose
- Sucrose + Hesperetin (Experimental): 7% (w/v) sucrose in water + 50 mg/L Hesperetin
  Interventions: Drug: Sucrose+ Hesperetin
- 7% sucrose (Experimental): 7% (w/v) sucrose in water
  Interventions: Other: 7% Sucrose

INTERVENTIONS:
Other: 10% Sucrose — 10% sucrose corresponding to a regular soft drink
  Other Names: table sugar
  Arms: 10% Sucrose
Drug: Sucrose+ Hesperetin — Addition of hesperetin increases sweetness of 7% sucrose solution to match sweetness of 10% sucrose solution
  Other Names: (2S)-3',5,7-Trihydroxy-4'-methoxyflavan-4-one; CAS number 520-33-2
  Arms: Sucrose + Hesperetin
Other: 7% Sucrose — 7% sucrose to match the caloric content of the sugar-reduced hesperetin intervention
  Other Names: table sugar
  Arms: 7% sucrose

SUMMARY:
The aim of this cross-over intervention study is to investigate the influence of hesperetin applied in combination with sucrose in comparison to an equally sweet-tasting sucrose-only solution and an isocaloric sucrose-only solution on markers of energy metabolism

DETAILED DESCRIPTION:
The study is designed as a randomised cross-over intervention study with three arms. The aim is to investigate the influence of a 10% sucrose solution, corresponding to the sugar content of a conventional soft drink, compared to an equally sweet-tasting 7% sucrose solution in combination with 50 mg/L of the polyphenol hesperetin, and a less sweet 7% sucrose solution w/o hesperetin on time-dependent blood glucose fluctuations and ad libitum energy intake in metabolically healthy male volunteers.

To investigate the underlying mechanisms, the individual appetite score, metabolic and hormonal responses to the interventions and will be measured. In addition, the participants' individual thresholds for sweet taste, preference and consumption for sweet-tasting foods such as sugar and sweeteners, and their body composition will be recorded as potential influencing factors.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoking
* normal taste responses towards sweet taste

Exclusion Criteria:

* pregnancy or breast-feeding
* regular smokers
* disturbed glucose and/or lipid metabolism
* regular intake of medication
* known allergies against one of the test compounds
* ageusia alcohol or drug addiction intake of antibiotics within the past 2 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2024-03-31 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose concentration | 15, 30, 60, 90, and 120 minutes after drinking the test solution
  Change compared to baseline in blood glucose concentration [mg/dL] in plasma samples after drinking the test solution
Change in appetite score | Difference between before and 120 minutes after drinking of the test solution
  Change compared to baseline in the subjective rating of the individual feeling of hunger, fullness, as well as appetite for a snack or for something sweet on a unstructured, digital visual analog scale ranging from 0-10 cm in comparison to baseline
Change in food intake | 120 minutes after drinking of the test solution
  Ad libitum food intake from a standardized breakfast

SECONDARY OUTCOMES:
Change in regulating hormones | 15, 30, 60, 90, and 120 minutes after drinking the test solution
  Change compared to baseline in Insulin, Glucagon-like peptide 1, Gastric inhibitory polypeptide, and Polypetide Y concentrations [mmol/L] in plasma samples after drinking the test solution

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lieder, PhD, Principal Investigator — University of Vienna
Locations (1):
- Christian Doppler Laboratory for Taste Research, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No